CLINICAL TRIAL: NCT04478552
Title: Randomized Controlled Trial on Analgesic Effect of Pre-operative Fascia Iliaca Compartment Block in Geriatric Patients With Hip Fracture
Brief Title: Analgesic Effect of Fascia Iliaca Compartment Block in Geriatric Patients With Hip Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United Christian Hospital (Other)
Responsible Party: Principal Investigator, Wan Tze Kit, Dr Wan Tze Kit, United Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPv1
Record Dates: First submitted 2020-03-25; First posted 2020-07-20 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Hip Fractures
Keywords: hip fracture; orthogeriatrics; fascia iliaca compartment block
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Procedure: Fascia iliaca compartment block
- Control group (Placebo Comparator)
  Interventions: Procedure: Placebo injection

INTERVENTIONS:
Procedure: Fascia iliaca compartment block — It involves injecting local anaesthetic agent (levobupivacaine) into the fascia iliaca compartment of the patient, infiltrating three major nerves that supply the medial, anterior and lateral thigh, namely the femoral and lateral femoral cutaneous nerves. This procedure can be done with anatomical landmark approach or under image guidance.
  Arms: Intervention group
Procedure: Placebo injection — same volume of normal saline, instead of levobupivacaine, will injected using the same technique.
  Arms: Control group

SUMMARY:
As population in Hong Kong is aging, incidence of geriatrics hip fractures rises. Operative treatment for selective patients offers pain control, early mobilization and reduction in medical morbidities and mortalities. Research has shown that the pain from hip fracture left untreated may have significant physical and psychological effects on the patient, precipitating delirium, especially in elderly patients with hip fractures, and may delay operative management and may complicate hospital stay. Studies report that the pain management for limb fractures in the elderly is hugely sub-optimal with some suggesting that only 2% receive adequate analgesia. Adequate analgesia before definitive treatment of hip fracture may improve mobilization and cognitive performance. As a part of multi-modal pain management, Fascia iliaca compartment block is being increasingly popular as a simple, safe and effective regional technique for patients with hip fractures and proximal femoral shaft fractures, providing consistent analgesic effect for hip fracture patients, irrespective of the performing doctor's experience. This study aims to provide high level local evidence of the effect and efficacy of the fascia iliaca compartment block in preoperative pain control for patients with hip fracture admitted to Orthopaedic and Traumatology ward in United Christian Hospital.

DETAILED DESCRIPTION:
This study is a randomized control, single blinded trial. It tests the hypothesis that fascia iliaca compartment block using local anaesthetic agent for pre-operative analgesia in patients with hip fracture, compared to that using normal saline as control, leads to a better pain control and fewer doses of systemic analgesics required. All patients admitted to United Christian Hospital Orthopaedic and Traumatology ward for hip fracture with radiological diagnosis will be seen by on-call resident. Principal investigator and other investigators will be notified of the admission within 1 working day. Subjects will be recruited according to inclusion and exclusion criteria as mentioned in the below section. Subjects will be recruited only if an informed consent for this study has been signed. Only patients with hip fracture pending emergency operation will be recruited. 2 enclosed envelopes will be prepared, in which one indicates "intervention", and one indicates "control". Subjects will randomly choose any of the envelopes without knowing the intervention/control group assignment. To maintain true randomization, the 2 envelopes will be kept in good condition, preventing identification of the underlying assignment from the outer appearance. Investigators, knowing the group assignment, will then prepare an injection kit set for Fascia iliaca compartment block which includes vials of levobupivacaine, normal saline, syringes, 22G/21G needle, simple dressing set and skin antiseptic solution. For the intervention group, fascia iliaca compartment block with 30ml/40ml 0.25% levobupivacaine, depending on body weight (30ml for body weight less than 50kg, 40ml for body weight more than 50kg), will be performed by investigators under landmark approach. For the control group, same volume of normal saline, instead of levobupivacaine, will injected using the same technique, so that single blinding can be achieved. Subjects' vital signs will be observed for every 10 minutes for 30 minutes after injection.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or above
* Patients admitted Orthopaedic and Traumatology ward in United Christian Hospital
* Radiographically confirmed unilateral fracture hip
* Patient requiring pre-operative analgesia
* Mentally competent
* Informed consent signed

Exclusion Criteria:

* Age less than 65
* Presence of more than one fracture
* Patient refusal to participating in this study
* Known true allergy or previous anaphylactic reaction to local anaesthetic
* Previous femoral-bypass surgery, or near a graft site.
* Previous surgery over the injection site
* Inflammation, infection, or hernia over the injection site
* INR >1.4
* Platelet count <100x 10^9/L
* Patient on heparin / fondaparinux / rivaroxaban / dabigatran / ticlopidine / clopidogrel / prasugrel / cilostazol

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Change in pain in terms of Numeric Rating Scale | on admission, just before fascia iliaca compartment block, 1 hour after injection, 12 hour after injection, 24 hour after injection, and 48 hour after injection.
  Numeric Rating Scale (0-10) whereas 0 is the least pain and 10 is the worst pain

CONTACTS AND LOCATIONS:
Locations (1):
- United Christian Hospital, Kwun Tong, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No